CLINICAL TRIAL: NCT01257113
Title: Is Supervised Exercise Therapy a Better Option Than Home Exercises for Patients With Subacromial Impingement When Looking at Pain and Function?
Brief Title: Supervised Exercise Therapy vs Home Exercises for Patients With Subacromial Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/2591
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder pain; shoulder impingement; rotatorcuff pathology; supervised exercise; homebased exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- supervised exercise (Experimental): The group gets 10 supervised exerciseclasses at the physiotherapy clinic in addition to homebased exercises
  Interventions: Other: supervised exercise
- homebased exercises (Experimental): The group gets 1 supervised exerciseclass before they do all their exercises at home
  Interventions: Other: homebased exercises

INTERVENTIONS:
Other: supervised exercise — This group will receive 10 classes of supervised exercise in the 6 weeks intervention. In this classes the patients will be with a physiotherapist that will adjust their home-exercise program and make sure they do the exercises in a good way. They will receive 4-6 exercises they shall do 3 times with 30 repetitions, 2 times every day. If necessary, they should also do stretching exercises
  Arms: supervised exercise
Other: homebased exercises — This group will receive 1 class of supervised exercise at the beginning of the 6 weeks intervention. In this class the patients will be with a physiotherapist that will put together a home-exercise program and make sure they do the exercises in a good way. They will receive 4-6 exercises they shall do 3 times with 30 repetitions, 2 times every day. If necessary, they should also do stretching exercises
  Arms: homebased exercises

SUMMARY:
The purpose of this study is to determine whether there are any difference between supervised exercise therapy and homebased exercise when looking at pain and function for patients with shoulder pain.

DETAILED DESCRIPTION:
Shoulder pain is common in the population. Various treatment modalities are used. According to the literature, it is equally good results for home exercises and for guided exercise therapy. The purpose of this study is to look at this again and determine whether there are any difference between supervised exercise therapy and homebased exercise when looking at pain and function for patients with subacromial impingement.

ELIGIBILITY:
Inclusion Criteria:

* Pain in one shoulder
* Had the condition for more than 12 weeks
* Pain at abduction (must be present in some part between 60 and 120 degrees)
* Pain/ weakness in isometric external rotation
* Positive Hawkins test

Exclusion Criteria:

* Instability
* Labral pathology
* Acromioclavicular joint (AC-joint) pathology
* Complete rupture in the rotatorcuff
* Glenohumeral osteoarthritis
* Previously operated on current shoulder
* The pain comes from neck pathology
* Rheumatoid arthritis or other serious physical or mental illness
* Lack of Norwegian language
* Unable to start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain and function 1 | Baseline
  Shoulder Pain and Disability Index
Pain and function 2 | At 6 weeks
  Shoulder Pain and Disability Index
Pain and function 3 | At 6 months
  Shoulder Pain and Disability Index

SECONDARY OUTCOMES:
Fear avoidance 1 | Baseline
  Fear-Avoidance Beliefs Questionnaire. Modified version with questions about shoulder instead of back
Fear avoidance 2 | At 6 weeks
  Fear-Avoidance Beliefs Questionnaire. Modified version with questions about shoulder instead of back.
Quality of life 1 | Baseline
  The Short-Form 36 questionnaire
Quality of life 2 | At 6 weeks
  The Short-Form 36 questionnaire
Pain the last week | Baseline and once a week for 6 weeks
  Numeric pain rating scale
Active range of motion 1 | Baseline
  Abduction, flexion, external rotation and internal rotation measured with inclinometer
Active range of motion 2 | At 6 weeks
  Abduction, flexion, external rotation and internal rotation measured with inclinometer
Impingement tests 1 | Baseline
  Hawkins test, painful arc test and isometric external rotation test is beeing conducted and scored positive or negative
Impingement tests 2 | At 6 weeks
  Hawkins test, painful arc test and isometric external rotation test is beeing conducted and scored positive or negative
Work status 1 | Baseline
  Registration of the patients work status
Work status 2 | At 6 weeks
  Registration of the patients work status
Work status 3 | At 6 months
  Registration of the patients work status
Patient satisfaction | At 6 weeks
  2 questions, one question about benefit and one about satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Ottar Vasseljen, Dr.Philos, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Tverrfaglig Poliklinikk, rygg-nakke-skulder. Fys.Med. og rehab., St.Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Granviken F, Vasseljen O. Home exercises and supervised exercises are similarly effective for people with subacromial impingement: a randomised trial. J Physiother. 2015 Jul;61(3):135-41. doi: 10.1016/j.jphys.2015.05.014. Epub 2015 Jun 18. PMID 26093810